CLINICAL TRIAL: NCT07362836
Title: Fruquintinib Versus Bevacizumab Plus Chemotherapy as Second-Line Therapy for Patients With RAS-Mutant Metastatic Colorectal Cancer (FRU-RAS): A Multicenter Randomized Controlled Trial
Brief Title: Fruquintinib Versus Bevacizumab Plus Chemotherapy in Second-Line RAS-Mutant Metastatic Colorectal Cancer (FRU-RAS)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C140
Record Dates: First submitted 2026-01-04; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fruquintinib+chemotherapy (Experimental): fruquintinib combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen)
  Interventions: Drug: fruquintinib+chemotherapy
- bevacizumab+chemotherapy (Active Comparator): bevacizumab combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen)
  Interventions: Drug: bevacizumab+chemotherapy

INTERVENTIONS:
Drug: fruquintinib+chemotherapy — fruquintinib combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen)
  Arms: fruquintinib+chemotherapy
Drug: bevacizumab+chemotherapy — bevacizumab combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen)
  Arms: bevacizumab+chemotherapy

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of fru+chemo as second-line therapy for patients with RAS-Mutant Metastatic Colorectal Cancer, especially when compared with the standard therapy BEV+chemo.

The trial aims to provide this kind of patients with a more beneficial therapeutic option.

Eligible patients were randomly assigned to the experimental group or the control group at a ratio of 1:1, Experimental group: Patients received fruquintinib combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen), Control group: Patients received bevacizumab combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen),

DETAILED DESCRIPTION:
Eligible patients were randomly assigned to the experimental group or the control group at a ratio of 1:1, stratified by bevacizumab treatment history (yes vs no), and metastatic sites (≤2 vs >2).

Experimental group: Patients received fruquintinib combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen), with the choice of oxaliplatin-based or irinotecan-based chemotherapy regimen depending on the previous chemotherapy regimen (chemotherapy switch): fruquintinib: 4mg, qd po, d1-21, q4w; FOLFIRI regimen: irinotecan 180mg/m2 intravenous infusion for 30-90min on days 1 and 15; LV 400mg/m2 intravenous infusion for 2h on days 1 and 15; 5-FU 400mg/m2 intravenous push on days 1 and 15, followed by 1200mg/(m2∙d) × 2d continuous intravenous infusion (total 2400mg/m2, infusion 46-48h); every 4 weeks as a treatment cycle. mFOLFOX6 regimen: oxaliplatin 85mg/m2 intravenous infusion for 2h on days 1 and 15; LV 400mg/m2 intravenous infusion for 2h on days 1 and 15; 5-FU 400mg/m2 intravenous push on days 1 and 15, followed by 1200mg/(m2∙d) × 2d continuous intravenous infusion (total 2400mg/m2, infusion 46-48h); every 4 weeks as a treatment cycle.

Control group: Patients received bevacizumab combined with chemotherapy (mFOLFOX6 or FOLFIRI regimen), with the choice of oxaliplatin-based or irinotecan-based chemotherapy regimen depending on the previous chemotherapy regimen (chemotherapy switch): bevacizumab: 5mg/kg, ivgtt, d1, 15, q4w; FOLFIRI regimen: irinotecan 180mg/m2 intravenous infusion for 30-90min on days 1 and 15; LV 400mg/m2 intravenous infusion for 2h on days 1 and 15; 5-FU 400mg/m2 intravenous push on days 1 and 15, followed by 1200mg/(m2∙d) × 2d continuous intravenous infusion (total 2400mg/m2, infusion 46-48h); every 4 weeks as a treatment cycle. mFOLFOX6 regimen: oxaliplatin 85mg/m2 intravenous infusion for 2h on days 1 and 15; LV 400mg/m2 intravenous infusion for 2h on days 1 and 15; 5-FU 400mg/m2 intravenous push on days 1 and 15, followed by 1200mg/(m2∙d) × 2d continuous intravenous infusion (total 2400mg/m2, infusion 46-48h); every 4 weeks as a treatment cycle.

During the combination treatment period, the tumor response was evaluated by imaging every 8 weeks. After at least 6 cycles of continuous administration, the following evaluations were made: ① If the patient met the conditions for conversion therapy, radical local treatments such as surgical resection or radiofrequency ablation could be performed. Patients in the fruquintinib group needed to discontinue the drug for about 2 weeks before surgery, while those in the bevacizumab group needed to discontinue for about 6 weeks. ② Patients who achieved disease control entered the maintenance treatment stage and received fruquintinib combined with chemotherapy or bevacizumab combined with chemotherapy, with the chemotherapy regimen determined by the doctor. The treatment continued until disease progression, intolerable toxicity, or withdrawal of informed consent occurred. During the maintenance treatment period, the tumor response was evaluated by imaging every 8 weeks. Safety observation indicators included adverse events, changes in laboratory indicators, vital signs, and electrocardiogram changes. The subsequent tumor treatment and survival follow-up after progression were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study, sign the informed consent form, and have good compliance.
2. 18 years ≤ age ≤ 75 years.
3. Histologically and/or cytologically confirmed unresectable metastatic colorectal cancer.
4. RAS mutant type.
5. Previously received chemotherapy based on fluoropyrimidines (5-fluorouracil or capecitabine, etc.), oxaliplatin or irinotecan; previous adjuvant/neoadjuvant therapy is allowed. If recurrence or metastasis occurs during or within 6 months after adjuvant/neoadjuvant therapy, it is considered as the failure of first-line systemic chemotherapy for advanced disease.
6. Patients must have at least one measurable lesion (RECIST 1.1).
7. ECOG performance status 0-1.
8. Expected survival ≥ 12 weeks.
9. Blood tests (without blood transfusion within 14 days) 1) Absolute neutrophil count ≥ 1.5×10^9/L, platelet count ≥ 100×10^9/L, hemoglobin concentration ≥ 9g/dL; 2) Liver function tests (AST and ALT ≤ 2.5×ULN, bilirubin ≤ 1.5×ULN; if there is liver metastasis, AST and ALT ≤ 5×ULN); 3) Renal function (serum creatinine (Cr) ≤ 1.5×ULN, or creatinine clearance rate (CCr) ≥ 60ml/min); 4) Coagulation, international normalized ratio (INR) ≤ 1.5×ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN; 5) Thyroid function, thyroid stimulating hormone (TSH) ≤ upper limit of normal (ULN); if abnormal, FT3 and FT4 levels should be examined, and patients with normal FT3 and FT4 levels can be included.
10. Women of childbearing age are willing to use medically approved effective contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study and for 3 months after the last administration of the study drug; for male subjects whose partners are of childbearing age, it is recommended to take effective contraceptive measures during the study and for 3 months after the last administration of the study drug.

Exclusion Criteria:

1. Enrolled in another clinical study within the 4 weeks prior to enrollment in this study;
2. Previously received anti-angiogenic small molecule targeted drug treatment, such as fruquintinib, etc.;
3. Symptomatic brain or leptomeningeal metastases (except for those who have undergone local radiotherapy or surgery for brain metastases for more than 6 months and have stable disease control);
4. Experienced severe infection within 4 weeks prior to enrollment (e.g., requiring intravenous infusion of antibiotics, antifungal drugs, or antiviral drugs);
5. Hypertension that cannot be well controlled with antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
6. Had active bleeding or coagulation disorders within 2 months prior to enrollment, had a bleeding tendency or was receiving thrombolytic therapy, and was assessed by the investigator as unsuitable for enrollment;
7. Had active heart disease within 6 months prior to treatment, including myocardial infarction, severe/unstable angina pectoris. Echocardiography showed left ventricular ejection fraction < 50%, or had poorly controlled arrhythmia;
8. Had other malignant tumors within 5 years prior to enrollment or at the same time (except for cured basal cell carcinoma of the skin and cervical carcinoma in situ);
9. Known to be allergic to the study drug or any of its excipients;
10. Unable to take oral medication or the investigator judged that the subject had a condition that affected drug absorption;
11. Pregnant (positive pregnancy test before medication) or breastfeeding women;
12. Had active or uncontrolled severe infections 1) Known human immunodeficiency virus (HIV) infection; 2) Known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must be excluded from active HBV infection, i.e., HBV DNA positive (>1×10^4 copies/mL or >2000 IU/mL); 3) Known hepatitis C virus (HCV) infection and HCV RNA positive (>1×10^3 copies/mL), or other hepatitis, liver cirrhosis;
13. Urinalysis indicated proteinuria ≥ 2+, and 24-hour urine protein quantification > 1.0g;
14. Other situations judged by the investigator as unsuitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-Free Survival (PFS) is a time-to-event outcome commonly used as a primary or secondary endpoint in oncology clinical trials. It quantifies the duration a patient lives without disease progression or death, providing an early indicator of treatment efficacy.

SECONDARY OUTCOMES:
Objective Response Rate | ORR will be assessed up to Week 24 after randomization
  ORR (Objective Response Rate) refers to the proportion of patients in a clinical trial whose tumor burden is reduced by a predefined amount, specifically achieving either a Complete Response (CR) or Partial Response (PR), as assessed by the investigator based on RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
Disease Control Rate | DCR will be assessed up to Week 24 after randomization.
  Disease Control Rate (DCR) is defined as the percentage of patients whose disease responds to treatment (i.e., achieves Complete Response (CR) or Partial Response (PR)) or remains stable (Stable Disease, SD) over a defined period of time. It reflects the proportion of patients who experience tumor shrinkage or disease stabilization without progression.
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 60 months
  Overall Survival (OS) is the most definitive and direct measure of clinical benefit in cancer trials. It is defined as the time from randomization (or start of treatment) to death from any cause. This endpoint captures the ultimate outcome of interest: whether a patient is alive.